CLINICAL TRIAL: NCT01177813
Title: A Phase III Randomised, Double-blind, Placebo-controlled Parallel Group Efficacy and Safety Study of BI 10773 and Sitagliptin Administered Orally Over 24 Weeks, in Drug naïve Patients With Type 2 Diabetes Mellitus and Insufficient Glycaemic Control Despite Diet and Exercise
Brief Title: Efficacy and Safety of Empagliflozin (BI 10773) Versus Placebo and Sitagliptin Over 24 Weeks in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1245.20; 2009-016243-20 (EudraCT Number: EudraCT)
Record Dates: First submitted 2010-07-29; First posted 2010-08-09 (Estimated); Results first posted 2014-06-16 (Estimated); Last update posted 2014-06-16 (Estimated); Status verified 2014-05

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin; Sitagliptin Phosphate

ARMS (5):
- BI 10773 low dose (Experimental): Patients receive BI 10773 low dose tablets once daily
  Interventions: Drug: Placebo identical to BI10773 high dose; Drug: BI 10773; Drug: Placebo identical to Sitagliptin 100mg
- BI 10773 high dose (Experimental): Patients receive BI 10773 high dose tablets once daily
  Interventions: Drug: Placebo identical to BI10773 low dose; Drug: BI10773; Drug: Placebo identical to Sitagliptin 100mg
- Placebo (Placebo Comparator): Patients receive tablets identical to those containing BI 10773 low dose and high dose and to Sitagliptin
  Interventions: Drug: Placebo identical to BI10773 low dose; Drug: Placebo identical to Sitagliptin 100mg; Drug: Placebo identical to BI10773 high dose
- Sitagliptin 100 mg (Active Comparator): Patients receive Sitagliptin 100 mg tablets once daily
  Interventions: Drug: Placebo identical to BI10773 high dose; Drug: Sitagliptin; Drug: Placebo identical to BI10773 low dose
- BI 10773 high dose open label (Experimental): Patients receive BI 10773 high dose tablets open label once daily
  Interventions: Drug: BI 10773 open label

INTERVENTIONS:
Drug: Placebo identical to BI10773 high dose — placebo tablets once daily
  Arms: BI 10773 low dose
Drug: BI 10773 — BI 10773 low dose tablet once daily
  Arms: BI 10773 low dose
Drug: BI 10773 open label — Patients receive BI 10773 high dose tablets open label once daily
  Arms: BI 10773 high dose open label
Drug: Placebo identical to BI10773 low dose — placebo tablets once daily
  Arms: BI 10773 high dose
Drug: Placebo identical to BI10773 low dose — placebo tablets once daily
  Arms: Placebo
Drug: Placebo identical to BI10773 high dose — placebo tablets once daily
  Arms: Sitagliptin 100 mg
Drug: Placebo identical to Sitagliptin 100mg — placebo tablets once daily
  Arms: Placebo
Drug: Placebo identical to Sitagliptin 100mg — placebo tablets once daily
  Arms: BI 10773 low dose
Drug: BI10773 — BI 10773 high dose tablets once daily
  Arms: BI 10773 high dose
Drug: Sitagliptin — Sitagliptin tablets 100 mg once daily
  Arms: Sitagliptin 100 mg
Drug: Placebo identical to Sitagliptin 100mg — placebo tablets once daily
  Arms: BI 10773 high dose
Drug: Placebo identical to BI10773 low dose — placebo tablets once daily
  Arms: Sitagliptin 100 mg
Drug: Placebo identical to BI10773 high dose — placebo tablets once daily
  Arms: Placebo

SUMMARY:
The aim of this study is to investigate the efficacy, safety and tolerability of BI 10773 compared to placebo and sitagliptin given for 24 weeks as monotherapy in patients with T2DM with insufficient glycaemic control. For the open-label part of the study the objective is to estimate the efficacy and safety of BI 10773 when given for 24 weeks in patients with T2DM with very poor glycaemic control.

ELIGIBILITY:
Inclusion criteria:

1. Diagnosis of type 2 diabetes mellitus prior to informed consent;
2. Male and female patients on diet and exercise regimen who are drug-naïve;
3. HbA1c >= 7.0% and <= 10.0% at Visit 1 (screening) for randomised treatment; HbA1c > 10.0% at visit 1 (screening) for the open-label BI 10773 arm;
4. Age >= 20 (Japan); Age >= 18 (countries other than Japan);
5. BMI <= 45 kg/m2 at Visit 1 (screening);
6. Signed and dated written informed consent by date of Visit 1

Exclusion criteria:

1. Uncontrolled hyperglycaemia;
2. Acute coronary syndrome (non-STEMI, STEMI and unstable angina pectoris), stroke or TIA within 3 months prior to informed consent;
3. Indication of liver disease, either ALT, AST, or alkaline phosphatase above 3 x ULN;
4. Impaired renal function (eGFR<50 ml/min);
5. Bariatric surgery within the past two years or other GI surgeries;
6. Medical history of cancer;
7. Contraindications to sitagliptin;
8. Blood dyscrasias or any disorders causing haemolysis or unstable red blood cell;
9. Treatment with any anti-diabetes drug within 12 weeks prior to randomisation;
10. Treatment with anti-obesity drugs or any other treatment leading to unstable body weight;
11. Current treatment with systemic steroids or change in dosage of thyroid hormones within 6 weeks prior to informed consent or any other uncontrolled endocrine disorder except T2DM;
12. Pre-menopausal women who are nursing or pregnant or are of child-bearing potential and not practicing an acceptable method of birth control;
13. Alcohol or drug abuse;
14. Intake of an investigational drug in another trial within 30 days prior to intake of study medication in this trial;
15. Any other clinical condition that would jeopardize patients safety while participating in this clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 986 (Actual)
Dates: Start 2010-07; Primary Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (124):
- United States (27):
  - 1245.20.10124 Boehringer Ingelheim Investigational Site, Mesa, Arizona
  - 1245.20.10108 Boehringer Ingelheim Investigational Site, Phoenix, Arizona
  - 1245.20.10150 Boehringer Ingelheim Investigational Site, Hot Springs, Arkansas
  - 1245.20.10154 Boehringer Ingelheim Investigational Site, Chino, California
  - 1245.20.10009 Boehringer Ingelheim Investigational Site, Santa Ana, California
  - 1245.20.10131 Boehringer Ingelheim Investigational Site, West Hills, California
  - 1245.20.10038 Boehringer Ingelheim Investigational Site, Northglenn, Colorado
  - 1245.20.10137 Boehringer Ingelheim Investigational Site, Clearwater, Florida
  - 1245.20.10006 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 1245.20.10085 Boehringer Ingelheim Investigational Site, Plantation, Florida
  - 1245.20.10078 Boehringer Ingelheim Investigational Site, Tampa, Florida
  - 1245.20.10080 Boehringer Ingelheim Investigational Site, Decatur, Georgia
  - 1245.20.10128 Boehringer Ingelheim Investigational Site, Avon, Indiana
  - 1245.20.10060 Boehringer Ingelheim Investigational Site, Fishers, Indiana
  - 1245.20.10065 Boehringer Ingelheim Investigational Site, Indianapolis, Indiana
  - 1245.20.10117 Boehringer Ingelheim Investigational Site, Arkansas City, Kansas
  - 1245.20.10039 Boehringer Ingelheim Investigational Site, Wichita, Kansas
  - 1245.20.10146 Boehringer Ingelheim Investigational Site, Louisville, Kentucky
  - 1245.20.10144 Boehringer Ingelheim Investigational Site, Watertown, Massachusetts
  - 1245.20.10115 Boehringer Ingelheim Investigational Site, Brick, New Jersey
  - 1245.20.10129 Boehringer Ingelheim Investigational Site, Carlisle, Ohio
  - 1245.20.10045 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 1245.20.10119 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 1245.20.10130 Boehringer Ingelheim Investigational Site, Gallipolis, Ohio
  - 1245.20.10089 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1245.20.10151 Boehringer Ingelheim Investigational Site, Hurst, Texas
  - 1245.20.10155 Boehringer Ingelheim Investigational Site, San Antonio, Texas
- Belgium (15):
  - 1245.20.32008 Boehringer Ingelheim Investigational Site, Brussels
  - 1245.20.32011 Boehringer Ingelheim Investigational Site, Brussels
  - 1245.20.32023 Boehringer Ingelheim Investigational Site, Brussels
  - 1245.20.32003 Boehringer Ingelheim Investigational Site, De Pinte
  - 1245.20.32015 Boehringer Ingelheim Investigational Site, Deurne
  - 1245.20.32016 Boehringer Ingelheim Investigational Site, Deurne
  - 1245.20.32025 Boehringer Ingelheim Investigational Site, Gozée
  - 1245.20.32022 Boehringer Ingelheim Investigational Site, Landen
  - 1245.20.32019 Boehringer Ingelheim Investigational Site, Leopoldsburg
  - 1245.20.32024 Boehringer Ingelheim Investigational Site, Linkebeek
  - 1245.20.32021 Boehringer Ingelheim Investigational Site, Mouscron
  - 1245.20.32027 Boehringer Ingelheim Investigational Site, Retie
  - 1245.20.32020 Boehringer Ingelheim Investigational Site, Sint-Gillis-Waas
  - 1245.20.32018 Boehringer Ingelheim Investigational Site, Tielt
  - 1245.20.32026 Boehringer Ingelheim Investigational Site, Tremelo
- Canada (19):
  - 1245.20.20011 Boehringer Ingelheim Investigational Site, Chilliwack, British Columbia
  - 1245.20.20018 Boehringer Ingelheim Investigational Site, Victoria, British Columbia
  - 1245.20.20015 Boehringer Ingelheim Investigational Site, Winnipeg, Manitoba
  - 1245.20.20012 Boehringer Ingelheim Investigational Site, Moncton, New Brunswick
  - 1245.20.20016 Boehringer Ingelheim Investigational Site, Mount Pearl, Newfoundland and Labrador
  - 1245.20.20008 Boehringer Ingelheim Investigational Site, St. John's, Newfoundland and Labrador
  - 1245.20.20001 Boehringer Ingelheim Investigational Site, Barrie, Ontario
  - 1245.20.20019 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 1245.20.20010 Boehringer Ingelheim Investigational Site, London, Ontario
  - 1245.20.20017 Boehringer Ingelheim Investigational Site, London, Ontario
  - 1245.20.20003 Boehringer Ingelheim Investigational Site, Markham, Ontario
  - 1245.20.20009 Boehringer Ingelheim Investigational Site, Newmarket, Ontario
  - 1245.20.20013 Boehringer Ingelheim Investigational Site, Ottawa, Ontario
  - 1245.20.20005 Boehringer Ingelheim Investigational Site, Strathroy, Ontario
  - 1245.20.20002 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1245.20.20006 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1245.20.20014 Boehringer Ingelheim Investigational Site, Charlottetown, Prince Edward Island
  - 1245.20.20007 Boehringer Ingelheim Investigational Site, Montague, Prince Edward Island
  - 1245.20.20021 Boehringer Ingelheim Investigational Site, Trois-Rivières, Quebec
- China (23):
  - 1245.20.86007 Boehringer Ingelheim Investigational Site, Beijing
  - 1245.20.86008 Boehringer Ingelheim Investigational Site, Beijing
  - 1245.20.86001 Boehringer Ingelheim Investigational Site, Guangzhou
  - 1245.20.86002 Boehringer Ingelheim Investigational Site, Guangzhou
  - 1245.20.86003 Boehringer Ingelheim Investigational Site, Guangzhou
  - 1245.20.86012 Boehringer Ingelheim Investigational Site, Guiyang
  - 1245.20.86020 Boehringer Ingelheim Investigational Site, Hangzhou
  - 1245.20.86049 Boehringer Ingelheim Investigational Site, Jinan
  - 1245.20.86018 Boehringer Ingelheim Investigational Site, Jingzhou
  - 1245.20.86019 Boehringer Ingelheim Investigational Site, Nanchang
  - 1245.20.86010 Boehringer Ingelheim Investigational Site, Nanjing
  - 1245.20.86043 Boehringer Ingelheim Investigational Site, Nanjing
  - 1245.20.86016 Boehringer Ingelheim Investigational Site, Qingdao
  - 1245.20.86004 Boehringer Ingelheim Investigational Site, Shanghai
  - 1245.20.86005 Boehringer Ingelheim Investigational Site, Shanghai
  - 1245.20.86006 Boehringer Ingelheim Investigational Site, Shanghai
  - 1245.20.86057 Boehringer Ingelheim Investigational Site, Shenyang
  - 1245.20.86017 Boehringer Ingelheim Investigational Site, Shiyan
  - 1245.20.86013 Boehringer Ingelheim Investigational Site, Suzhou
  - 1245.20.86015 Boehringer Ingelheim Investigational Site, Taiyuan
  - 1245.20.86009 Boehringer Ingelheim Investigational Site, Wuhan
  - 1245.20.86011 Boehringer Ingelheim Investigational Site, Xi'an
  - 1245.20.86014 Boehringer Ingelheim Investigational Site, Xiamen
- Germany (11):
  - 1245.20.49013 Boehringer Ingelheim Investigational Site, Dresden
  - 1245.20.49016 Boehringer Ingelheim Investigational Site, Düsseldorf
  - 1245.20.49015 Boehringer Ingelheim Investigational Site, Frankfurt
  - 1245.20.49019 Boehringer Ingelheim Investigational Site, Haag
  - 1245.20.49020 Boehringer Ingelheim Investigational Site, Hohenmölsen
  - 1245.20.49014 Boehringer Ingelheim Investigational Site, Köthen
  - 1245.20.49002 Boehringer Ingelheim Investigational Site, Neuwied
  - 1245.20.49008 Boehringer Ingelheim Investigational Site, Nuremberg
  - 1245.20.49017 Boehringer Ingelheim Investigational Site, Saint Ingbert/Oberwürzbach
  - 1245.20.49022 Boehringer Ingelheim Investigational Site, Schauenburg
  - 1245.20.49003 Boehringer Ingelheim Investigational Site, Unterschneidheim
- India (10):
  - 1245.20.91005 Boehringer Ingelheim Investigational Site, Bangalore
  - 1245.20.91006 Boehringer Ingelheim Investigational Site, Bangalore
  - 1245.20.91008 Boehringer Ingelheim Investigational Site, Bangalore
  - 1245.20.91003 Boehringer Ingelheim Investigational Site, Belagavi
  - 1245.20.91004 Boehringer Ingelheim Investigational Site, Chennai
  - 1245.20.91009 Boehringer Ingelheim Investigational Site, Chennai
  - 1245.20.91002 Boehringer Ingelheim Investigational Site, Mumbai
  - 1245.20.91007 Boehringer Ingelheim Investigational Site, Mumbai, Maharastra
  - 1245.20.91010 Boehringer Ingelheim Investigational Site, Nagpur
  - 1245.20.91001 Boehringer Ingelheim Investigational Site, Tamil Nadu
- Ireland (5):
  - 1245.20.35302 Boehringer Ingelheim Investigational Site, Co. Cork
  - 1245.20.35305 Boehringer Ingelheim Investigational Site, Co. Galway
  - 1245.20.35303 Boehringer Ingelheim Investigational Site, Co. Wexford
  - 1245.20.35304 Boehringer Ingelheim Investigational Site, Offaly
  - 1245.20.35306 Boehringer Ingelheim Investigational Site, Wexford
- Japan (12):
  - 1245.20.81007 Boehringer Ingelheim Investigational Site, Chiyoda-ku, Tokyo
  - 1245.20.81001 Boehringer Ingelheim Investigational Site, Chuo-ku, Tokyo
  - 1245.20.81002 Boehringer Ingelheim Investigational Site, Chuo-ku, Tokyo
  - 1245.20.81005 Boehringer Ingelheim Investigational Site, Ebetsu, Hokkaido
  - 1245.20.81004 Boehringer Ingelheim Investigational Site, Kamakura, Kanagawa
  - 1245.20.81003 Boehringer Ingelheim Investigational Site, Minato-ku, Tokyo
  - 1245.20.81006 Boehringer Ingelheim Investigational Site, Shinjuku-ku, Tokyo
  - 1245.20.81008 Boehringer Ingelheim Investigational Site, Shinjuku-ku, Tokyo
  - 1245.20.81009 Boehringer Ingelheim Investigational Site, Suita, Osaka
  - 1245.20.81010 Boehringer Ingelheim Investigational Site, Ube, Yamaguchi
  - 1245.20.81012 Boehringer Ingelheim Investigational Site, Urasoe, Okinawa
  - 1245.20.81013 Boehringer Ingelheim Investigational Site, Urasoe, Okinawa
- Switzerland (2):
  - 1245.20.41004 Boehringer Ingelheim Investigational Site, Lugano
  - 1245.20.41003 Boehringer Ingelheim Investigational Site, Rorschach

REFERENCES:
- [Derived] Natale P, Tunnicliffe DJ, Toyama T, Palmer SC, Saglimbene VM, Ruospo M, Gargano L, Stallone G, Gesualdo L, Strippoli GF. Sodium-glucose co-transporter protein 2 (SGLT2) inhibitors for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 May 21;5(5):CD015588. doi: 10.1002/14651858.CD015588.pub2. PMID 38770818
- [Derived] Tuttle KR, Levin A, Nangaku M, Kadowaki T, Agarwal R, Hauske SJ, Elsasser A, Ritter I, Steubl D, Wanner C, Wheeler DC. Safety of Empagliflozin in Patients With Type 2 Diabetes and Chronic Kidney Disease: Pooled Analysis of Placebo-Controlled Clinical Trials. Diabetes Care. 2022 Jun 2;45(6):1445-1452. doi: 10.2337/dc21-2034. PMID 35472672
- [Derived] Cherney D, Lund SS, Perkins BA, Groop PH, Cooper ME, Kaspers S, Pfarr E, Woerle HJ, von Eynatten M. The effect of sodium glucose cotransporter 2 inhibition with empagliflozin on microalbuminuria and macroalbuminuria in patients with type 2 diabetes. Diabetologia. 2016 Sep;59(9):1860-70. doi: 10.1007/s00125-016-4008-2. Epub 2016 Jun 17. PMID 27316632
- [Derived] Roden M, Weng J, Eilbracht J, Delafont B, Kim G, Woerle HJ, Broedl UC; EMPA-REG MONO trial investigators. Empagliflozin monotherapy with sitagliptin as an active comparator in patients with type 2 diabetes: a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Diabetes Endocrinol. 2013 Nov;1(3):208-19. doi: 10.1016/S2213-8587(13)70084-6. Epub 2013 Sep 9. PMID 24622369

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Patients receive tablets identical to those containing 10 mg and 25 mg Empagliflozin and to Sitagliptin 100 mg once daily in the morning.
- Empagliflozin10 mg: Patients receive 10 mg Empagliflozin in tablets once daily in the morning.
- Empagliflozin 25 mg: Patients receive 25 mg Empagliflozin in tablets once daily in the morning.
- Sitagliptin 100 mg: Patients receive 100 mg Sitagliptin in tablets once daily in the morning.
- Empagliflozin 25 mg OL: Patients receive 25 mg Empagliflozin in tablets open label (OL) once daily in the morning.
Period: Overall Study
Arm/Group | Placebo | Empagliflozin10 mg | Empagliflozin 25 mg | Sitagliptin 100 mg | Empagliflozin 25 mg OL
Started | 228 | 224 | 224 | 223 | 87
Completed | 187 | 206 | 204 | 206 | 78
Not Completed | 41 | 18 | 20 | 17 | 9
Not completed — Adverse Event | 8 | 2 | 4 | 6 | 3
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 3 | 2 | 2 | 0 | 1
Not completed — Lost to Follow-up | 12 | 5 | 6 | 3 | 0
Not completed — Withdrawal by Subject | 12 | 7 | 6 | 5 | 3
Not completed — Other reason not defined above | 5 | 2 | 2 | 3 | 2

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) including all randomised and treated patients who had a baseline HbA1c value (non-open label groups) and Open-label set including all patients entered in the empagliflozin 25 mg open-label treatment arm.
Groups:
- Sitagliptin 100: Patients receive 100 mg Sitagliptin in tablets once daily in the morning.
- Empagliflozin 25 mg OL: Patients receive 25 mg Empagliflozin in tablets open label once daily in the morning.
- Total: Total of all reporting groups
Arm/Group | Placebo | Empagliflozin10 mg | Empagliflozin 25 mg | Sitagliptin 100 | Empagliflozin 25 mg OL | Total
Number analyzed (Participants) | 228 | 224 | 224 | 223 | 87 | 986
Age, Continuous [Mean (Standard Deviation); unit: years] — The descriptive statistics for Total refers to the 4 non-open label groups (Placebo, Empagliflozin 10mg and 25 mg, Sitagliptin)
  years | 54.9 (10.9) | 56.2 (11.6) | 53.8 (11.6) | 55.1 (9.9) | 50.2 (11.3) | 55.0 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 82 | 79 | 82 | 23 | 371
  Male | 123 | 142 | 145 | 141 | 64 | 615

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Haemoglobin (HbA1c) After 24 Weeks
Description: The term "baseline" refers to the last observation before the start of randomised trial treatment (or of open-label treatment for the open-label arm).
  In this endpoint, the "measured values" show unadjusted values, whereas the statistical analyses show adjusted values. Statistics for open-label group are descriptive.
Time Frame: Baseline and day 169
Population: FAS and open-label set, last observation carried forward (LOCF) was used as the imputation rule for both sets
Measure: Mean (Standard Error); unit: percent of HbA1c
Arm/Group | Placebo | Empagliflozin10 mg | Empagliflozin 25 mg | Sitagliptin 100 mg | Empagliflozin 25 mg OL
Number analyzed (Participants) | 228 | 224 | 224 | 223 | 87
percent of HbA1c | 0.06 (0.05) | -0.66 (0.06) | -0.77 (0.06) | -0.65 (0.05) | -3.10 (0.22)
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin10 mg; Model was adjusted for treatment,geographical region, and renal function at baseline as fixed effects, and baseline HbA1c as linear covariate; Test type: Superiority or Other; p < 0.0001, ANCOVA — Difference calculated as empagliflozin 10mg minus placebo; Mean Difference (Final Values) = -0.74, 97.5% CI 2-sided [-0.90 to -0.57], Standard Error of Mean 0.07
Statistical Analysis 2: Comparison: Placebo vs Empagliflozin 25 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — Difference calculated as empagliflozin 25mg minus placebo; Mean Difference (Final Values) = -0.85, 97.5% CI 2-sided [-1.01 to -0.69], Standard Error of Mean 0.07

2. Secondary Outcome: Change From Baseline to Week 24 in Body Weight
Description: as for outcome 1
Time Frame: Baseline and day 169
Population: FAS (LOCF) and open-label set (LOCF)
Measure: Mean (Standard Error); unit: kg
Arm/Group | Placebo | Empagliflozin10 mg | Empagliflozin 25 mg | Sitagliptin 100 mg | Empagliflozin 25 mg OL
Number analyzed (Participants) | 228 | 224 | 224 | 223 | 87
kg | -0.33 (0.15) | -2.26 (0.19) | -2.48 (0.18) | 0.17 (0.18) | -1.93 (0.44)
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin10 mg; Model was adjusted for treatment,geographical region,and renal function at baseline as fixed effects,baseline body weight and baseline HbA1c as linear covariate; Test type: Superiority or Other; p < 0.0001, ANCOVA — Difference calculated as empagliflozin 10mg minus placebo; Mean Difference (Final Values) = -1.93, 97.5% CI 2-sided [-2.48 to -1.38], Standard Error of Mean 0.24
Statistical Analysis 2: Comparison: Placebo vs Empagliflozin 25 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — Difference calculated as empagliflozin 25mg minus placebo; Mean Difference (Final Values) = -2.15, 95% CI 2-sided [-2.70 to -1.60], Standard Error of Mean 0.24

3. Secondary Outcome: Change From Baseline to Week 24 in Systolic and Diastolic Blood Pressure (SBP and DBP)
Description: The term "baseline" refers to the last observation before the start of randomised trial treatment (or of open-label treatment for the open-label arm).
  In this endpoint, the "measured values" show unadjusted values, whereas the statistical analyses show adjusted values. Statistics for open-label group are descriptive.
  For blood pressure, data following changes in antihypertensive therapy is censored, in the same way that data following initiation of rescue medication is censored.
Time Frame: Baseline and week 24
Population: FAS and open-label set, last observation carried forward without values following a change in antihypertensive therapy (LOCF- H) was used as the imputation rule
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Empagliflozin10 mg | Empagliflozin 25 mg | Sitagliptin 100 mg | Empagliflozin 25 mg OL
Number analyzed (Participants) | 228 | 224 | 224 | 223 | 87
mmHg
  Systolic blood pressure | 0.0 (0.8) | -3.5 (1.0) | -3.2 (0.9) | 0.2 (0.9) | -3.8 (1.2)
  Diastolic blood pressure | -0.4 (0.5) | -1.1 (0.6) | -1.7 (0.5) | 0.4 (0.5) | -1.5 (0.8)
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin10 mg; Comparison for Systolic Blood Pressure Model was adjusted for treatment,geographical region, and renal function at baseline as fixed effects, baseline SBP and baseline HbA1c as linear covariate; Test type: Superiority or Other; p = 0.0231, ANCOVA — Difference calculated as empagliflozin 10mg minus placebo; Mean Difference (Final Values) = -2.6, 97.5% CI 2-sided [-5.2 to 0.0], Standard Error of Mean 1.1
Statistical Analysis 2: Comparison: Placebo vs Empagliflozin 25 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0028, ANCOVA — Difference calculated as empagliflozin 25mg minus placebo; Mean Difference (Final Values) = -3.4, 97.5% CI 2-sided [-6.0 to -0.9], Standard Error of Mean 1.1
Statistical Analysis 3: Comparison: Placebo vs Empagliflozin10 mg; Comparison for diastolic blood pressure Model was adjusted for treatment,geographical region, and renal function at baseline as fixed effects, baseline DBP and baseline HbA1c as linear covariate; Test type: Superiority or Other; p = 0.3987, ANCOVA — Difference calculated as empagliflozin 10mg minus placebo; Mean Difference (Final Values) = -0.6, 97.5% CI 2-sided [-2.1 to 0.9], Standard Error of Mean 0.7
Statistical Analysis 4: Comparison: Placebo vs Empagliflozin 25 mg; [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; p = 0.0296, ANCOVA — Difference calculated as empagliflozin 25mg minus placebo; Mean Difference (Final Values) = -1.5, 97.5% CI 2-sided [-3.0 to 0.0], Standard Error of Mean 0.7

4. Other Pre Specified Outcome: Confirmed Hypoglycaemic Adverse Events
Description: Confirmed hypoglycaemic events refer to all hypoglycaemic events, that had a glucose value <= 70 ml/dL or where assistance was required.
  Symptomatic hypoglycaemic events were to be reported as adverse events. Patients can be counted in more than one category.
Time Frame: From first drug intake until 7 days after last medication intake, up to 219 days
Population: Treated set (actual) including all patients treated with at least 1 dose of randomised trial medication with some treatment switchers (1 from Empa25 to placebo; 1 patient got Empa 10 at least with one mis-allocated kit) and open-label set
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Empagliflozin10 mg | Empagliflozin 25 mg | Sitagliptin 100 mg | Empagliflozin 25 mg OL
Number analyzed (Participants) | 229 | 224 | 223 | 223 | 87
percentage of participants
  Symptomatic hypoglycaemic adverse events | 0.4 | 0.4 | 0.4 | 0.4 | 0
  Asymptomatic hypoglycaemic adverse events | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From first drug administration until seven days after last trial medication intake, up to 219 days
Arm/Group | Placebo | Empagliflozin10 mg | Empagliflozin 25 mg | Sitagliptin 100 mg | Empagliflozin 25 mg OL
Serious Adverse Events (participants affected / at risk) | 6/229 | 8/224 | 5/223 | 6/223 | 3/87
Other Adverse Events (participants affected / at risk) | 63/229 | 45/224 | 36/223 | 44/223 | 27/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=229) | Empagliflozin10 mg (N=224) | Empagliflozin 25 mg (N=223) | Sitagliptin 100 mg (N=223) | Empagliflozin 25 mg OL (N=87)
Herpes virus infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Goitre (Endocrine disorders) | 0 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Diabetic neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Vertebrobasilar insufficiency (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 1 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Colonic polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 1 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Breast mass (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Gilbert's syndrome (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0
Hernia (General disorders) | 0 | 0 | 0 | 1 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Animal bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=229) | Empagliflozin10 mg (N=224) | Empagliflozin 25 mg (N=223) | Sitagliptin 100 mg (N=223) | Empagliflozin 25 mg OL (N=87)
Nasopharyngitis (Infections and infestations) | 17 | 16 | 11 | 15 | 1
Urinary tract infection (Infections and infestations) | 9 | 14 | 8 | 11 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 35 | 5 | 4 | 13 | 14
Dyslipidaemia (Metabolism and nutrition disorders) | 10 | 13 | 10 | 6 | 7
Diarrhoea (Gastrointestinal disorders) | 3 | 4 | 3 | 3 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.